CLINICAL TRIAL: NCT05364710
Title: Clinical Poof-of-concept Study on Rapid Immune Modulating Effects
Brief Title: Clinical Proof-of-concept Study on Rapid Immune Modulating Effects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 058-006
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Immune Surveillance

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blinded, cross-over study design.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will not be informed on which intervention they receive on any given day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Crossover study: Participants will be consuming placebo on a clinic day at least 1 week prior to a clinic day where he/she will consume the active intervention.
  Interventions: Dietary Supplement: Transfer factor from colostrum ultrafiltrate
- Group B (Experimental): Crossover study: Participants will be consuming the active intervention on a clinic day at least 1 week prior to a clinic day where he/she will consume placebo.
  Interventions: Dietary Supplement: Transfer factor from colostrum ultrafiltrate

INTERVENTIONS:
Dietary Supplement: Transfer factor from colostrum ultrafiltrate — Proteins that confer immune protection, isolated from cow colostrum ultrafiltrate and used to promote immune health and surveillance.

SUMMARY:
Clinical-proof-of concept study, comparing the acute immune impacts of of 2 doses of a novel blend of supplements to a placebo. This study involves twenty-four participants, composed of healthy adults, who will be taking a placebo and 2 different doses of the blend at different times. Testing for immune status and cytokine levels will be conducted to determine the acute impact of the blend on immune function as compared to the placebo.

DETAILED DESCRIPTION:
Clinical-proof-of-concept study comparing the acute immune effects of 2 doses of a nutraceutical blend, and a placebo. The nutraceutical blend is based on a transfer factor isolated from cow colostrum ultrafiltrate.

24 subjects will participate in a placebo-controlled, randomized, double-blinded, cross-over study design, wherein they will be taking placebo, dose 1, and dose 2, each separated by a 1-week washout period.

Blood samples are taken 1 hour after participants arrive; the dose is then administered. Samples are taken 1 hour, 2 hours, and 24 hours following administration. At each blood sample collection, a spit sample will also be taken for salivary IgA testing.

A series of immune panels will be used to determine the acute impacts on immune surveillance, immune cell activation status, immune cell priming, and cytokine profiles.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Veins easy to see in one or both arms
* Willing to comply with study procedures, including
* Maintaining a consistent diet and lifestyle routine throughout the study;
* Consistent habit of bland breakfast on days of clinic visits
* Abstaining from exercising on and nutritional supplements on the morning of a study visit;
* Abstaining from use of coffee, tea, and soft drinks for at least one hour prior to a clinic visit;
* Abstaining from music, candy, gum, computer/cell phone use, during clinic visits

Exclusion Criteria:

* Previous major gastrointestinal surgery
* Taking anti-inflammatory medications on a daily basis
* Currently experiencing intense stressful events/life changes
* Currently in intensive athletic training (such as marathon runner)
* Currently taking antipsychotic medications such as clozapine, Risperdal, Abilify, Zyprexa or Seroquel
* An unusual sleep routine
* Unwilling to maintain a constant intake of supplements over the duration of the study
* Anxiety about having blood drawn
* People of childbearing potential: Pregnant, nursing, or trying to become pregnant
* Known food sensitivities related to ingredients in active test product placebo Prescription medication evaluated on a cas-by-case basis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-05-07 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Immune communication | 2 hours
  Observation of changes in serum cytokine levels

SECONDARY OUTCOMES:
Immune Surveillance and Alertness | 2 hours
  Observation of changes in immune cell trafficking and status of immune cell alertness, ie. the changes in immune cell populations and activation following administration.

OTHER OUTCOMES:
Immune responsiveness | 2 hours
  Ex vivo immune challenges, observing the capabilities of anti-bacterial and anti-viral defenses. Additionally, mucosal immune protection as determined by salivary IgA, defensins, and transferrin changes.

CONTACTS AND LOCATIONS:
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No